CLINICAL TRIAL: NCT02052518
Title: Early Childhood Obesity Prevention Program: Building Better Families and Communities
Brief Title: Early Childhood Obesity Prevention Program
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: University of Connecticut (Other); UConn Health (Other)
Responsible Party: Principal Investigator, Michelle Cloutier, MD, Professor of Pediatrics, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HD073966-02
Record Dates: First submitted 2014-01-27; First posted 2014-02-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Body Weight Changes
Keywords: Childhood obesity; Breastfeeding; Introduction of solids; Introduction of juice
MeSH Terms: conditions — Body Weight Changes; Pediatric Obesity; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced NFN Home Program (Experimental): Education and Skill set training with materials to implement the behaviors recommended. Using a motivational interviewing framework, intervention participants will receive dietary and activity counseling, develop a Family Wellness Plan and will be linked to community resources.
  Interventions: Behavioral: Experimental
- Nurturing Family Network Home Visitation (Placebo Comparator): Mothers will receive the standard of care from the Nurturing Families Network Home Visitation program
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — These participants will receive the enhanced intervention including decision support and problem solving skills in addition to the standard of care for the individuals in the Nuturing Family Network Home Visition Program
  Other Names: Enhanced NFN Home Program

SUMMARY:
This study is proposed on behalf of the Hartford Childhood Wellness Alliance, a 107 member, 35 group organization whose goal is to improve the health of children in Hartford, CT. In a randomized control trial, the primary aim of this study is to test the initial efficacy of a program of enhanced home visitation with neighborhood and community support to change maternal behaviors related to infant nutrition (sweetened beverage/juice consumption, breastfeeding and introduction of solids), parenting skills (establishing routines around sleep, reading cues for hunger, satiety, television time) and family wellness (improving the home food environment, enhancing physical activity). The investigators hypothesize that at 12 months of age, infants in the intervention arm will drink less sugar sweetened beverages/juices, will have ingested solids at an older age, will have been breastfed longer and more exclusively than infants in the control arm and will have less TV viewing, more established sleep routines and greater soothability (primary outcomes).

DETAILED DESCRIPTION:
See Manuscript: 125. Cloutier MM, Wiley J, Wang Z, Grant A, Gorin AA. The Early Childhood Obesity Prevention Program (ECHO): An ecologically-based intervention delivered by home visitors for newborns and their mothers. BMC Public Health, 15:584 PMID 26073106, 2015.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Nurturing Families Network Program
* Singleton birth >34 weeks gestation
* Any race or ethnicity
* ECHO neighborhood
* Mothers and their newborns

Exclusion Criteria:

* Mothers or newborns with special health care needs
* Infant with major malformation
* Small for Gestational Age/low birth weight

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of months of breast feeding | 6 and 12 months
  Number of months that child is breastfed

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Cloutier, MD, Principal Investigator — Connecticut Children's Medical Centr
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
When final analysis has been completed and manuscripts have been published, data will be made available upon request to other investigators

REFERENCES:
- [Derived] Cloutier MM, Wiley J, Wang Z, Grant A, Gorin AA. The Early Childhood Obesity Prevention Program (ECHO): an ecologically-based intervention delivered by home visitors for newborns and their mothers. BMC Public Health. 2015 Jun 24;15:584. doi: 10.1186/s12889-015-1897-9. PMID 26104068